CLINICAL TRIAL: NCT00817687
Title: A Randomised, Multicenter, Open-label Study Evaluating the Impact on the Fibrosis at Week 52 of an Early Biopsy at (D10) Versus Standard Management in Patients Who Have Undergone de Novo Renal Transplantation and Received a Marginal Organ Transplant
Brief Title: A Study of the Impact of an Early Biopsy in Patients Treated With CellCept (Mycophenolate Mofetil) After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21655
Record Dates: First submitted 2008-12-16; First posted 2009-01-06 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]
- 2 (No Intervention)
  Interventions: Drug: mycophenolate mofetil [CellCept]

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept] — As prescribed; + early biopsy
  Arms: 1
Drug: mycophenolate mofetil [CellCept] — As prescribed; + standard treatment
  Arms: 2

SUMMARY:
This 2 arm study will evaluate the impact on fibrosis at week 52 of an early biopsy, in patients who have received a kidney transplant from an expanded criteria donor. Patients will be randomized to one of two groups; the first group will have a biopsy at day 10, and the second group will receive standard management. All patients will be given CellCept as standard of care. The anticipated time on study treatment is 1 year, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* in receipt of an initial cadaveric kidney transplant;
* in receipt of graft with biopsy;
* in receipt of a 'marginal' kidney transplant.

Exclusion Criteria:

* in receipt of a second kidney transplant;
* in receipt of a multi-organ transplant or a double kidney transplant;
* malignant tumor, or a history of cancer in past 5 years, other than successfully treated basal cell or spinocellular cancer or cancer in situ of cervix;
* replicating hepatitis B and/or C, or HIV positive serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with >=25% increase in fibrosis score | Day 0 to Week 52

SECONDARY OUTCOMES:
Renal function (creatinine clearance) | From randomization to Week 52
Incidence and time of occurrence of clinical acute rejection | From randomization to Week 52
Adverse events, laboratory parameters, cancers and lymphoproliferative syndromes | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- France (16):
  - Besançon
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - Lille
  - Limoges
  - Marseille
  - Nantes
  - Paris
  - Poitiers
  - Rouen
  - Salouël
  - Strasbourg
  - Suresnes
  - Tours
  - Vandœuvre-lès-Nancy